CLINICAL TRIAL: NCT06750614
Title: Systematic Assessment of the Modulatory Role of Brain State on the Prefrontal Response to Excitatory Stimulation: a Concurrent RTMS/fNIRS Pilot Study
Brief Title: Exploring the Modulatory Role of Brain State on the Prefrontal Response to Excitatory Stimulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Georg Kranz, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HSEARS20230324002
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Healthy Adult
Keywords: Intermittent Theta-burst Stimulation, iTBS; Brain State; Transcranial Magnetic Stimulation, TMS; Functional Near-infrared Spectroscopy (fNIRS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mood (Active Comparator): During concurrent iTBS/fNIRS, stimuli with positive, negative, and neutral valence will be presented to participants to induce the corresponding mood.
  Interventions: Device: intermittent theta-burst stimulation (iTBS)
- Cognitive Task (Active Comparator): During concurrent iTBS/fNIRS, the effects of participants' cognitive load will be assessed by performing the backward counting task.
  Interventions: Device: intermittent theta-burst stimulation (iTBS)
- Relax (Active Comparator): During concurrent iTBS/fNIRS, participants will be instructed to relax.
  Interventions: Device: intermittent theta-burst stimulation (iTBS)

INTERVENTIONS:
Device: intermittent theta-burst stimulation (iTBS) — In each visit, the intensity of the iTBS applied to the participant will be set at 70% of their individual resting motor threshold (rMT), with one session specifically targeting the left DLPFC.

SUMMARY:
Therapeutic repetitive transcranial magnetic stimulation (rTMS) for depression is well-supported, with multiple protocols approved by the United States Food and Drug Administration and global efforts aimed at boosting its antidepressant effects underway. However, there exists an under-reported aspect of clinical trials using rTMS: what are patients doing during each stimulation session? Here, the investigators begin this investigation with individuals without a history of depression nor other psychiatric diagnosis. The investigators focus on the underlying brain activity. The investigators will systematically assess the modulatory role of brain state on the brain's response to a session of rTMS by using a concurrent, non-invasive brain imaging setting: functional near-infrared spectroscopy (fNIRS), marking the first effort of its kind in this field.

DETAILED DESCRIPTION:
The scientific literature on rTMS rehabilitation is steadily growing and new treatment protocols that aim to optimize rehabilitation efficacy as well as efficiency are emerging. However, no consideration to what patients should be doing during rTMS treatment sessions is given. These details are typically omitted in the literature, and advice is not given in recent guidelines. When details are reported, patients are assumed to enter a relaxed state during treatment. This assumption is highly problematic, especially for MDD because depression is an internalizing disorder, wherein emotional and cognitive dyscontrol are major features linked with abnormal activity of the dorsolateral prefrontal cortex (DLPFC), the region being stimulated. Indeed, instructing patients to concentrate on thoughts that exacerbate their depressive symptoms during stimulation diminishes the antidepressant treatment effect, and cognitive neuroscience research suggests the importance of considering the initial brain state when conducting behavioral and neuroimaging experiments with TMS. Attention to what occurs during stimulation is highly relevant but usually omitted in neuropsychiatric rehabilitation research. This proposal is a systematic assessment of the modulatory role of brain state on the prefrontal response to rTMS in healthy participants. Results from this study will inform whether the clinical literature on therapeutic rTMS is mistaken for not controlling for brain state, and provide proof-of-concept for future clinical trials and collaborative research proposals (CRF) for the treatment of neuropsychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* Biological and mental health, based on a clinical interview
* Able to understand and follow instructions

Exclusion Criteria:

* Major internal diseases, neurological disorders, or mental disorders
* Having a metal implant
* Hearing problems or in-ear ringing
* Pregnancy or breastfeeding
* Any conditions that will contraindicate to iTBS or fNIRS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Oxygenated hemoglobin (HbO) change | Through study completion, an average of 1 year
  iTBS-induced HbO change in the DLPFC measured by fNIRS

SECONDARY OUTCOMES:
Deoxygenated hemoglobin (HbR) change | Through study completion, an average of 1 year
  iTBS-induced HbR change in the DLPFC measured by fNIRS

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No